CLINICAL TRIAL: NCT04845178
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase 2 Study of ABP-450 (prabotulinumtoxinA) Purified Neurotoxin Complex for the Prevention of Migraine Headache
Brief Title: Investigation of Safety and Efficacy of ABP-450 for Migraine Prevention in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEON Biopharma, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABP-20001
Record Dates: First submitted 2021-03-28; First posted 2021-04-14 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — prabotulinumtoxin A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Approximately 765 patients will be randomized in a 1:1:1 ratio and receive 1 of the following 3 treatments: ABP-450 Low Dose, ABP-450 High Dose, or placebo via intramuscular injection into pre-specified areas of the head and neck.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator, study nurse/other study personnel, and patients will be blinded to the treatment group. An appropriately trained person will reconstitute investigational product, fill masked-labeled syringes and provide them to the investigator, but will not perform any assessments with the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABP-450 - Low Dose (Experimental): ABP-450 Low Dose - intramuscular injections into specified muscles.
  Interventions: Drug: ABP-450
- ABP-450 - High Dose (Experimental): ABP-450 High Dose - intramuscular injections into specified muscles.
  Interventions: Drug: ABP-450
- Placebo (Placebo Comparator): Placebo (0.9% saline, sterile, unpreserved, USP/Ph.Eur) intramuscular injections into specified muscles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABP-450 — ABP-450 (prabotulinumtoxinA) contains a 900 kDa botulinum toxin type-A complex produced by the bacterium Clostridium botulinum.
  Other Names: prabotulinumtoxinA
  Arms: ABP-450 - High Dose; ABP-450 - Low Dose
Drug: Placebo — 0.9% sodium chloride, sterile, unpreserved, USP/PhEur
  Other Names: 0.9% sodium chloride; saline
  Arms: Placebo

SUMMARY:
This Phase 2 trial will evaluate the efficacy and safety of ABP-450 for migraine prevention in adults who suffer from six or more migraine days per month. The study will enroll 765 patients across approximately 64 sites in the United States, Canada and Australia. Study subjects will be divided evenly across a low dose group, a high dose group and a placebo group. All patients will receive two treatment cycles of ABP-450 or placebo utilizing the Company's novel injection paradigm.

DETAILED DESCRIPTION:
The Phase 2 trial will evaluate the efficacy and safety of ABP-450 for migraine prevention in adults who suffer from six or more migraine days per month. The study will enroll 765 patients across approximately 64 sites in the United States, Canada and Australia. Study subjects will be divided evenly across a low dose of ABP-450 group, a high dose of ABP-450 group, and a placebo group. All patients will receive two treatment cycles utilizing the Company's novel treatment paradigm involving fewer injections than the current botulinum toxin treatment option for chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Patient can understand the ICF, provides signed ICF and patient privacy information (eg, Authorization for Use and Release of Health and Research Study Information) before initiating any study-specific procedure, and agrees to comply with protocol requirements.
2. Male or female patients 18 years or older of age (no upper age limit) at the time of signing the informed consent.
3. Patient has at least a 1-year history of episodic migraine (with or without aura) or chronic migraine (with or without aura) according to the ICHD-3 (2018) definition and diagnostic criteria.
4. Age of the patient at the time of migraine onset <50 years.
5. History of, on average ≥6 migraine or probable migraine days per month in the 3 months prior to Screening.
6. Patient is on a stable dose of medications, if any, as recommended by the patient's health care practitioner, used for acute treatment of migraine for at least 3 months prior to Screening. Patient is not taking any migraine prophylactic treatment prohibited per protocol or if on prophylactic treatment has washed out.
7. A Woman of Child Bearing Potential (WOCBP) must be willing and able to use a medically acceptable and effective method of birth control as determined by the investigator, during the entire study.
8. A WOCBP must have a negative pregnancy test at Screening.
9. Patient is able to read, understand, and complete the eDiary.
10. Patient is willing and able to adhere to the study assessments, visit schedules, and prohibitions, as described in this protocol.

Exclusion Criteria:

Medical Conditions

1. History of migraine accompanied by diplopia or decreased level of consciousness, or retinal migraine.
2. Current diagnosis of chronic tension-type headache, new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or cranial neuropathy.
3. Confounding and clinically significant pain syndromes (eg, fibromyalgia, chronic low back pain, complex regional pain syndromes) as evaluated by the investigator.
4. Diagnosis of myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease that might interfere with the study.
5. Psychiatric conditions that are uncontrolled and/or untreated, including conditions that are not controlled for a minimum of 6 months prior to Screening as evaluated by the investigator. Patients with a lifetime history of psychosis, mania, or dementia are excluded.
6. History of addiction, including alcohol or drugs of abuse, within 6 months prior to Screening.
7. Hepatitis B (HBsAg positive) or hepatitis C (ie, detectable HCV RNA) virus infection.

   Note: Patients with a prior history of treated hepatitis B virus infection who are antigen negative or patients with a prior history of treated HCV infection who are HCV RNA undetectable may be considered after consultation with the study medical monitor.
8. Any infection or clinically significant skin problem in any of the injection sites.
9. Have been injected with anesthesia or steroids in the targeted muscles during the 30 days immediately prior to initiation of the Baseline period.
10. Any medical condition (including but not limited to viral or other active infections) that, in the opinion of the investigator, classifies the patient as unsuitable for participation in the study or patients who do not seem to be in good general health at the time of Screening, and prior to any investigational study drug administration.

    Note: Patients will not routinely be tested for COVID-19 during the study. Patients presenting with fever or who are symptomatic for COVID-19 will be required to be tested and treated through their general practitioner.

    Other Diagnostic Assessments
11. Significant risk of self-harm based on clinical interview and responses on the C-SSRS, or of harm to others in the opinion of the investigator; patients must be excluded if they report suicidal ideation with intent, with or without a plan (ie, Type 4 or 5 on the C-SSRS) in the past 6 months or report suicidal behavior in the past 6 months prior to Screening.
12. Body mass index ≥38 kg/m2 at Screening.

    Prior/Concomitant Medications and Treatments
13. Use of opioids or barbiturates >2 days per month in the 3 months prior to Screening.
14. Use of CBD or other types of cannabinoids in the 3 months prior to Screening and throughout the study.
15. Any use of botulinum toxin for migraine or any other medical reasons within 4 months prior to Screening and during the Screening and Baseline periods and at or above the shoulders at any time during the study.
16. Any monoclonal antibody CGRP inhibitor treatment (within or outside of a clinical study) within 6 months prior to Screening and throughout the study.
17. Any orally administered non-peptide CGRP antagonists (within or outside of a clinical study) within 4 weeks prior to the Baseline period and throughout the study.
18. Use of devices for the treatment of migraine (ie, non-invasive neuromodulation therapies including but not limited to non-invasive nerve stimulation [gammaCore], transcranial magnetic stimulation [Cefaly], external trigeminal nerve stimulation, transcutaneous electrical nerve stimulation, and peripheral neuroelectrical stimulation) during Screening and throughout the study.
19. Any other treatments or therapies (eg, acupuncture in head and neck region, cranial traction, nociceptive trigeminal inhibition, occipital nerve block treatments, and dental splints for headache) to the head, neck, or shoulder regions during Screening and throughout the study that, in the opinion of the investigator, would interfere with the investigational study drug.
20. History of inadequate response to 3 classes of medications (which have different mechanisms of action) prescribed for the prevention of migraine, excluding CGRP therapies.
21. History of hypersensitivity to human serum albumin, sucrose, or botulinum toxin type A or a positive test for botulinum toxin type A antibody.

    Prior/Concurrent Clinical Study Experience
22. Participation in another interventional study within 6 months prior to Screening and throughout the study.
23. Female patients planning on becoming pregnant during the course of the study and/or lactating/breastfeeding.
24. Patient has donated or lost a significant volume (>450 mL) of blood or plasma within 30 days of screening.
25. Patient is an employee or family member of the investigator, study site personnel, PPD, or AEON.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Change in Monthly Migraine Days | Baseline to Weeks 21 to 24 Treatment period.
  The primary efficacy endpoint will be the change in mean Monthly Migraine Days (MMD) from the 4-week Baseline period to Weeks 21 to 24 Treatment period.
Incidence of Treatment Emergent Adverse Events | Baseline to Week 28 - End of Study.
  The primary safety endpoint will be the incidence of TEAEs throughout the study when dosed with placebo, ABP-450 (low dose), or ABP-450 (high dose).

SECONDARY OUTCOMES:
Percentage of Patients with Reduction in Mean Migraine Days (MMD) | Baseline to Week 28 - End of Study.
  Percentage of patients with a reduction from Baseline of ≥ 50 percent, ≥ 75 percent and 100% percent in average number of MMD will be assessed by Treatment Group.
Mean change in Monthly Migraine Days (MMD) | Baseline to Week 28 - End of Study.
  Overall mean change from Baseline in the number of MMD will be assessed by Treatment Group.
Mean change in Monthly Migraine Days (MMD) requiring medications for acute treatment of migraine or headaches | Baseline to Week 28 - End of Study.
  Overall mean change from Baseline in number of MMD requiring migraine specific medication and non-specific medications for the acute treatment of migraine or headache will be assessed by Treatment Group.
Mean change in Headache Hours | Baseline to Week 28 - End of Study.
  Overall mean change from Baseline in headache (either moderate or severe) hours will be assessed by Treatment Group.
Mean Change in Monthly Headache Days | Baseline to Week 28 - End of Study.
  Overall mean change from Baseline in monthly headache days will be assessed by Treatment Group.
Mean change of Migraine-Specific-Quality of Life (MSQ) Domains | Baseline to Week 28 - End of Study.
  The Mean Change in Migraine-Specific-Quality of Life (MSQ), a 14-item assessment, with each item rated on a 6-point scale (ranging from "none of the time" to "all of the time") with higher scores indicating better quality of life will be assessed by Treatment Group.
Percentage of Patients with Reduction in Migraine Physical Function Impact Diary (MPFID) | Baseline to Week 28 - End of Study.
  Percentage of patients with a reduction from Baseline in the impact on Migraine Physical Function Impact Diary (MPFID) will be assessed by Treatment Group.
Suicidality by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to Week 28 - End of Study.
  Percentage of patients with Suicidal Ideation and Behaviors will be assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS).
Development of Anti-Drug Antibodies (ADA) to ABP-450 | Baseline to Week 28 - End of Study.
  Percentage of patients developing Anti-Drug Antibodies to ABP-450 antibodies (binding and if positive, neutralizing) will be assessed.

OTHER OUTCOMES:
Mean Change in Patient Global Impression of Change (PGI-C) Score | Baseline to Week 28 - End of Study.
  The Mean change in the subject's assessment of the change in clinical status since the start of treatment measured by the Patients' Global Impression of Change (PGI-C) Scale will be assessed by Treatment Group.
Mean Change in Patient Global Impression of Severity (PGI-S) Score | Baseline to Week 28 - End of Study.
  The Mean change in the subject's assessment of the severity of their condition since the start of treatment measured by the Patients' Global Impression of Severity (PGI-S) Scale will be assessed by Treatment Group.
Mean Change in MIgraine Disability Assessment Score (MIDAS) Total Score | Baseline to Week 28 - End of Study.
  The Mean Change in the Migraine Disability Assessment Scale (MIDAS) between Baseline and End of Treatment assessed by Treatment Group. MIDAS is a 5-item self-administered questionnaire. The 5 items sum to a total MIDAS score of 0 to 155. A higher score indicates greater headache-related disability (worse score).
Percentage of Patients with Reduction in the Physical Impairment Domaine Score of the Migraine Physical Function Impact Diary (MPFID) | Baseline to Week 28 - End of Study.
  Percentage of patients with a reduction from Baseline on Physical Impairment Domain Score measured by Migraine Physical Function Impact Diary (MPFID) assessed by Treatment Group.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Lipton, MD, Principal Investigator — Albert Einstein College of Medicine; Stewart J Tepper, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (62):
- United States (54):
  - MDFirst Research, Chandler, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Arizona Neuroscience Research, Phoenix, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Axiom Research LLC, Colton, California
  - Velocity Research San Diego, La Mesa, California
  - Collaborative Neuroscience Research, Long Beach, California
  - Los Angeles Headache Center, Los Angeles, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute For Clinical Research LLC - San Diego - ClinEdge - PPDS, San Diego, California
  - Delta Waves LLC - Hunt - PPDS, Colorado Springs, Colorado
  - Paradigm Clinical Research Centers, Wheat Ridge, Colorado
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Quality Research of South Florida, Hialeah, Florida
  - Sandhill Research, LLC, Lake Mary, Florida
  - Canvas Clinical Research, Lake Worth, Florida
  - BioMed Research Institute, INC, Miami, Florida
  - Medical Research Center, LLC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Clinical Research of Central Florida - ClinEdge - PPDS, Winter Haven, Florida
  - NeuroTrials Research Inc. - Clinedge - PPDS, Atlanta, Georgia
  - Drug Studies America, Inc, Marietta, Georgia
  - Velocity Clinical Research - Boise - ERN - PPDS, Meridian, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Kansas Institute of Research, LLC, Overland Park, Kansas
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - MedVadis Research, Waltham, Massachusetts
  - Quest Research Institute - Hunt - PPDS, Farmington Hills, Michigan
  - Henry Ford Allegiance Neurology, Jackson, Michigan
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Barrett Clinic, P.C. - Clinedge - PPDS, La Vista, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Wake Research - CRCN, LLC, Las Vegas, Nevada
  - Hassman Research Institute - ClinEdge - PPDS, Berlin, New Jersey
  - Albuquerque Clinical Trials Inc, Albuquerque, New Mexico
  - Dent Neurologic Institute, Amherst, New York
  - New York Neurology Associates, New York, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Centricity Research Dublin Multispecialty, Dublin, Ohio
  - The Orthopedic Foundation, New Albany, Ohio
  - Thomas Jefferson University, Jefferson Headache Center, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - WR-ClinSearch, Chattanooga, Tennessee
  - Bryant Research Group, Nashville, Tennessee
  - DCT - Baxter LLC dba Discovery Clinical Trials, Dallas, Texas
  - Mercury Clinical Research Incorporated, Sugar Land, Texas
  - Aspen Clinical Research LLC - Clinedge - PPDS, Orem, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Grampians Health, Ballarat, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Canada (4):
  - CARe Clinic, Red Deer, Alberta
  - True North Clinical Research, Halifax, Nova Scotia
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Diex Recherche Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data collected during the trial, after deidentification may be shared following review of the clinical study report by the FDA review division and if a decision is made to publish the results in an publication outside posting the results in clinicaltrials.gov